CLINICAL TRIAL: NCT03048292
Title: Reducing Disparities in Mechanical Embolectomy Access for Patients of New York City Via a Mobile Interventional Stroke Team: Systems of Care and Time-To-Treatment
Brief Title: New York City Mobile Interventional Stroke Team
Acronym: NYC MIST
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 16-1290
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Acute Stroke
Keywords: Embolectomy; Embolus; Thrombectomy; Thrombolysis; Thrombus; Mobile; Interventional; Neurointervention; Stroke; Ischemic; Acute; Endovascular; Cerebrovascular; Clot; Stent Retriever; Tissue Plasminogen Activator; Drip and Ship; Mothership; Trip and Treat
MeSH Terms: conditions — Stroke; Embolism; Thrombosis; Ischemia | interventions — Solitaire composite resin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Clot; Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Mobilized Neurointervention Team: Patients undergoing endovascular stroke interventions.
  Interventions: Other: Acute Endovascular Stroke Treatment
- Mobilized Patient
  Interventions: Other: Acute Endovascular Stroke Treatment
- Core Comprehensive Stroke Center Treatment
  Interventions: Other: Acute Endovascular Stroke Treatment

INTERVENTIONS:
Other: Acute Endovascular Stroke Treatment
  Other Names: Solitaire; Trevo; Embotrap; Medtronic; Stryker; Neuravi; Penumbra; Microvention

SUMMARY:
Endovascular treatment has recently become the recommended therapy for acute stroke after the publication of five randomized trials (MR CLEAN1, ESCAPE2, EXTEND IA3, SWIFT PRIME4, REVASCAT5) in 2015 that demonstrate its efficacy. Hospitals need to adapt to these updated stroke care guidelines, and many hospitals are not appropriately equipped for neurointerventional procedures. Decreased time to treatment is associated with favorable clinical outcomes, and best practices to optimize workflow between comprehensive stroke centers and secondary hospitals have become an important area of study. This prospective study is being conducted on acute stroke cases within the Mount Sinai Health System from 1 June 2016 up until 31 December 2018. The researchers would like to evaluate how variable methods of interventional service delivery for acute stroke affect clinical measures and outcomes.

More specifically, the researchers are conducting this study in order to determine whether outcomes of neurointervention for large vessel occlusion in stroke, for patients presenting to and receiving treatment at a comprehensive stroke center, will be superior to that delivered by a mobilized intervention team at a central satellite hospital. In particular, the hypothesis is that factors affecting outcome include presentation to secondary hospital, delays with transfer including traffic conditions and time of day, and the acquisition of complex imaging within secondary hospitals.

ELIGIBILITY:
Inclusion criteria:

- all patients who consent to the study and present with acute stroke treated with thrombectomy in the Mount Sinai Health System (Mount Sinai, Mount Sinai West, Mount Sinai Beth Israel, Mount Sinai St. Luke's) from 1 June 2016 - 31 December 2018.

Exclusion criteria:

* If the patient is pregnant
* Under age 18
* A prisoner. If timing of treatment cannot be captured, patients with these data points will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who consent to the study and present with acute stroke treated with thrombectomy in the Mount Sinai Health System.
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2016-06; Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Treatment times | 90 days
  Time between first hospital arrival and final recanalization

SECONDARY OUTCOMES:
Time to groin puncture procedure | 3 months
  Time of first hospital arrival to groin puncture
Time of EMS contact to groin puncture | 90 days
NIHSS | 90 days
  National Institutes of Health Stroke Scale (NIHSS) a 11-item impairment scale to evaluate neurologic outcome and degree of recovery.
  Each item is scored between 0 and up to 4, (0 normal function with higher score indicating higher level of impairment. with minimum score 0 and maximum possible score 42.
modified Rankin Scale (mRS) | 90 days
  the mRS measures degree of disability/dependence after a stroke. the mRS is a scale that runs from 0 (no symptoms) to 6 (death).

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Fifi, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (4):
- United States (4):
  - Mount Sinai Beth Israel, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai St Luke's, New York, New York
  - Mount Sinai Health System, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berkhemer OA, Fransen PS, Beumer D, van den Berg LA, Lingsma HF, Yoo AJ, Schonewille WJ, Vos JA, Nederkoorn PJ, Wermer MJ, van Walderveen MA, Staals J, Hofmeijer J, van Oostayen JA, Lycklama a Nijeholt GJ, Boiten J, Brouwer PA, Emmer BJ, de Bruijn SF, van Dijk LC, Kappelle LJ, Lo RH, van Dijk EJ, de Vries J, de Kort PL, van Rooij WJ, van den Berg JS, van Hasselt BA, Aerden LA, Dallinga RJ, Visser MC, Bot JC, Vroomen PC, Eshghi O, Schreuder TH, Heijboer RJ, Keizer K, Tielbeek AV, den Hertog HM, Gerrits DG, van den Berg-Vos RM, Karas GB, Steyerberg EW, Flach HZ, Marquering HA, Sprengers ME, Jenniskens SF, Beenen LF, van den Berg R, Koudstaal PJ, van Zwam WH, Roos YB, van der Lugt A, van Oostenbrugge RJ, Majoie CB, Dippel DW; MR CLEAN Investigators. A randomized trial of intraarterial treatment for acute ischemic stroke. N Engl J Med. 2015 Jan 1;372(1):11-20. doi: 10.1056/NEJMoa1411587. Epub 2014 Dec 17. PMID 25517348
- [Background] Goyal M, Demchuk AM, Menon BK, Eesa M, Rempel JL, Thornton J, Roy D, Jovin TG, Willinsky RA, Sapkota BL, Dowlatshahi D, Frei DF, Kamal NR, Montanera WJ, Poppe AY, Ryckborst KJ, Silver FL, Shuaib A, Tampieri D, Williams D, Bang OY, Baxter BW, Burns PA, Choe H, Heo JH, Holmstedt CA, Jankowitz B, Kelly M, Linares G, Mandzia JL, Shankar J, Sohn SI, Swartz RH, Barber PA, Coutts SB, Smith EE, Morrish WF, Weill A, Subramaniam S, Mitha AP, Wong JH, Lowerison MW, Sajobi TT, Hill MD; ESCAPE Trial Investigators. Randomized assessment of rapid endovascular treatment of ischemic stroke. N Engl J Med. 2015 Mar 12;372(11):1019-30. doi: 10.1056/NEJMoa1414905. Epub 2015 Feb 11. PMID 25671798
- [Background] Campbell BC, Mitchell PJ, Kleinig TJ, Dewey HM, Churilov L, Yassi N, Yan B, Dowling RJ, Parsons MW, Oxley TJ, Wu TY, Brooks M, Simpson MA, Miteff F, Levi CR, Krause M, Harrington TJ, Faulder KC, Steinfort BS, Priglinger M, Ang T, Scroop R, Barber PA, McGuinness B, Wijeratne T, Phan TG, Chong W, Chandra RV, Bladin CF, Badve M, Rice H, de Villiers L, Ma H, Desmond PM, Donnan GA, Davis SM; EXTEND-IA Investigators. Endovascular therapy for ischemic stroke with perfusion-imaging selection. N Engl J Med. 2015 Mar 12;372(11):1009-18. doi: 10.1056/NEJMoa1414792. Epub 2015 Feb 11. PMID 25671797
- [Background] Saver JL, Goyal M, Bonafe A, Diener HC, Levy EI, Pereira VM, Albers GW, Cognard C, Cohen DJ, Hacke W, Jansen O, Jovin TG, Mattle HP, Nogueira RG, Siddiqui AH, Yavagal DR, Baxter BW, Devlin TG, Lopes DK, Reddy VK, du Mesnil de Rochemont R, Singer OC, Jahan R; SWIFT PRIME Investigators. Stent-retriever thrombectomy after intravenous t-PA vs. t-PA alone in stroke. N Engl J Med. 2015 Jun 11;372(24):2285-95. doi: 10.1056/NEJMoa1415061. Epub 2015 Apr 17. PMID 25882376
- [Background] Jovin TG, Chamorro A, Cobo E, de Miquel MA, Molina CA, Rovira A, San Roman L, Serena J, Abilleira S, Ribo M, Millan M, Urra X, Cardona P, Lopez-Cancio E, Tomasello A, Castano C, Blasco J, Aja L, Dorado L, Quesada H, Rubiera M, Hernandez-Perez M, Goyal M, Demchuk AM, von Kummer R, Gallofre M, Davalos A; REVASCAT Trial Investigators. Thrombectomy within 8 hours after symptom onset in ischemic stroke. N Engl J Med. 2015 Jun 11;372(24):2296-306. doi: 10.1056/NEJMoa1503780. Epub 2015 Apr 17. PMID 25882510
- [Derived] Morey JR, Zhang X, Marayati NF, Matsoukas S, Fiano E, Oxley T, Dangayach N, Stein LK, Fara MG, Skliut M, Kellner C, De Leacy R, Mocco J, Tuhrim S, Fifi JT. Mobile Interventional Stroke Teams Improve Outcomes in the Early Time Window for Large Vessel Occlusion Stroke. Stroke. 2021 Aug;52(9):e527-e530. doi: 10.1161/STROKEAHA.121.034222. Epub 2021 Aug 5. PMID 34348472
- [Derived] Morey JR, Oxley TJ, Wei D, Kellner CP, Dangayach NS, Stein L, Hom D, Wheelwright D, Rubenstein L, Skliut M, Shoirah H, De Leacy RA, Singh IP, Zhang X, Persaud S, Tuhrim S, Dhamoon M, Bederson J, Mocco J, Fifi JT; Mount Sinai Stroke Investigators*. Mobile Interventional Stroke Team Model Improves Early Outcomes in Large Vessel Occlusion Stroke: The NYC MIST Trial. Stroke. 2020 Dec;51(12):3495-3503. doi: 10.1161/STROKEAHA.120.030248. Epub 2020 Nov 2. PMID 33131426